CLINICAL TRIAL: NCT03987789
Title: Intraoperative Protective Mechanical Ventilation in Patients Requiring Emergency Abdominal Surgery: IMPROVE-2 Multicenter Prospective Randomized Trial
Brief Title: Intraoperative Protective Mechanical Ventilation in Patients Requiring Emergency Abdominal Surgery
Acronym: IMPROVE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPROVE-2 study; 2019-A00265-52 (Other: ANSM)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-07

CONDITIONS: Emergency Abdominal Surgery; Mechanical Ventilation; General Anesthesia; Postoperative Morbidity
Keywords: Mechanical Ventilation; Lung-Protective Ventilation; Postoperative Pulmonary Complications; Postoperative morbidity

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, stratified, parallel-group clinical trial with blinded outcome assessment and concealed allocation of patients undergoing emergency abdominal surgery using low VT lung-protective ventilation to a strategy of minimal alveolar distension using low PEEP level or to a strategy aimed at increasing alveolar recruitment (higher PEEP level individually titrated to minimize the driving pressure in addition to recruitment maneuvers)
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to mask the assigned ventilation strategy from the treating clinicians because they have an ethical responsibility to ensure patient safety during the emergency procedures. However, procedures will be put in place to minimize the possibility of bias arising because research staff becomes aware of trial group allocation. At each participating center, patients will be followed up for primary and secondary endpoints by members of the research staff who will be unaware of the trial group allocation. Information on whether the primary and secondary outcomes occur will be collected and entered into the electronic web-based case report form (eCRF) by trial or clinical trained personal (clinical research associate), blinded to the allocation group, under the supervision of the local principal investigator (PI) or designee who will also be unaware of the trial group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low PEEP group (Active Comparator): Patients will receive a PEEP level ≤5 cmH2O without recruitment maneuvers
  Interventions: Other: Low PEEP
- Driving-pressure-guided group (Experimental): Patients will receive PEEP levels individually set at the highest possible value (up to 15 cmH2O) providing a driving pressure (airway plateau pressure minus PEEP) lower than 13 cmH2O, in addition to recruitment maneuvers
  Interventions: Other: Driving-pressure-guided group

INTERVENTIONS:
Other: Driving-pressure-guided group — Patients will receive PEEP levels individually set at the highest possible value (up to 15 cmH2O) providing a driving pressure (airway plateau pressure minus PEEP) lower than 13 cmH2O, in addition to recruitment maneuvers.
  Arms: Driving-pressure-guided group
Other: Low PEEP — Patients will receive a PEEP level ≤5 cmH2O without recruitment maneuvers
  Arms: Low PEEP group

SUMMARY:
The aim of this study is to compare the effects of a strategy aimed at increasing alveolar recruitment (high PEEP levels adjusted according to driving pressure and recruitment maneuvers) with that of a strategy aimed at minimizing alveolar distension (low PEEP level without recruitment maneuver) on postoperative respiratory failure and mortality in patients receiving low VT ventilation during emergency abdominal surgery.

DETAILED DESCRIPTION:
Emergency abdominal surgery is associated with a high risk of morbidity and mortality. Postoperative pulmonary complications (PPCs) are the second most common surgical complication and adversely influence surgical morbidity. Postoperative respiratory failure (PRF) is one of the most serious pulmonary complication.

Two hypotheses can be forward by the literature. First, a low VT lung protective ventilation in combination with a strategy aimed at minimizing alveolar distension by using low PEEP level (and without recruitment maneuver) could improve postoperative outcome while reducing the risk of hemodynamic alterations or, second, could increase the risk of PRF compared with a strategy aimed at increasing alveolar recruitment using higher PEEP level adjusted according to driving pressure in combination with recruitment maneuvers in adult patients undergoing emergency abdominal surgery. Given the uncertainties, and in order to determine the impact of lung protective ventilation strategies on clinical outcomes of high-risk surgical patients, a randomized trial is needed.

Our primary hypothesis is that, during low VT ventilation, a strategy aimed at increasing alveolar recruitment by using high PEEP levels adjusted according to driving pressure in combination with recruitment maneuvers could be more effective at reducing PRF and mortality after emergency abdominal surgery than a strategy aimed at minimizing alveolar distension by using lower PEEP without recruitment maneuver.

Given the number of patients for whom the question applies, the prevalence and the burden of PPCs, the study can have significant clinical importance and public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Patients requiring emergency (defined by the need to proceed to surgery within a few hours after diagnosis)
* Laparoscopic or non-laparoscopic abdominal surgery under general anesthesia and with an expected duration of at least two hours

Exclusion Criteria:

* Patients already receiving mechanical ventilation for more than 12 hours before enrollment
* Intracranial hypertension
* Chronic respiratory disease requiring oxygen therapy or mechanical ventilation at home
* Undrained pneumothorax or subcutaneous emphysema
* Patients for which death is deemed imminent and inevitable or patients with an underlying disease process with a life expectancy of less than 3 month
* Body mass index (BMI) >40 kg/m2
* Pregnant or breastfeeding women
* Patients already enrolled in the IMPROVE-2 trial
* Participation in a confounding trial with mortality or PRF as the main endpoint
* Patient's or relative's refusal to participate
* Guardianship or trusteeship patient
* No affiliation to the Social Security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Postoperative respiratory failure | Hospital discharge - Up to day 30
  Composite criteria :
  1. - Failure to wean from the ventilator after surgery (Yes or No)
  2. - Requiring unplanned reintubation (Yes or No)
  3. - Curative non-invasive ventilation once extubated postoperatively (Yes or No)
  4. - Death (all cause of mortality) (Yes or No)
  If at least one of these 4 criteria is answered yes, the composite criterion (i.e. the primary outcome) will be answered yes

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Day 30
  Hypoxemia, pneumonia? development of acute respiratory distress syndrome (ARDS)
Postoperative extra-pulmonary complications | Day 30
  sepsis and septic shock, renal dysfunction
SOFA | Day 1
  Sequential-related Organ Failure Assessment
SOFA | Day 2
  Sequential-related Organ Failure Assessment
SOFA | Day 3
  Sequential-related Organ Failure Assessment
SOFA | Day 4
  Sequential-related Organ Failure Assessment
SOFA | Day 5
  Sequential-related Organ Failure Assessment
SOFA | Day 6
  Sequential-related Organ Failure Assessment
SOFA | Day 7
  Sequential-related Organ Failure Assessment
Ventilator-free days | Day 30
  The number of days alive and with unassisted breathing
Duration of invasive mechanical ventilation | Up to Day 30
  Duration of invasive mechanical ventilation from randomization to first tracheal extubation
Total duration of mechanical ventilation | Up to Day 30
  Total duration of mechanical ventilation (additive, for all épisodes)
Time to successful tracheal extubation | 48 hours
  Absence of ventilatory support during the first 48 hours after extubation
Total volume of intraoperative fluids | Day 1
  Total volume of intraoperative fluids (crystalloids and colloids)
Median norepinephrine doses during surgery | Day 1
  µg/kg/min
Median phenylephrine doses during surgery | Day 1
  µg/kg/min
Median ephedrine doses during surgery | Day 1
  µg/kg/min
Intensive care unit (ICU)-free days | Day 30
  Intensive care unit (ICU)-free days
Duration of ICU stay | Up to day 90
  Duration of ICU stay
Duration of hospital stay | Up to day 90
  Duration of hospital stay
All-cause mortality | Day 30
  All-cause mortality
All-cause mortality | Day 90
  All-cause mortality
Time to death | Up to 90 days
  Time to death (Days)
Hemodynamic instability | Up to day 30
  Hemodynamic instability ventilatory-related defined as a drop of arterial systolic pressure below 80 mmHg for more than 5 minutes not responding to treatment
Pneumothorax | Up to day 30
  Pneumothorax ventilatory-related

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Futier, Principal Investigator — CHU de Clermont-Ferrand
Locations (28):
- France (28):
  - University hospital, Angers
  - Hospital, Annecy
  - University hospital, Besançon
  - University Hospital, Bordeaux
  - Hospital, Chalon-sur-Saône
  - University hospital, Clermont-Ferrand
  - University hospital, Dijon
  - University hospital, Grenoble
  - University hospital, Le Mans
  - University hospital, Lille
  - University hospital, Lyon
  - University hospital, Marseile
  - Assistance Publique-Hôpitaux de Marseille, Marseille
  - Institut Paoli Calmette, Marseille
  - University hospital, Marseille
  - University hospital, Montpellier
  - University Hospital, Nantes
  - University hospital, Nice
  - University hospital, Nîmes
  - Assistance Publique-Hôpitaux de Paris, Paris
  - Hospital, Périgueux
  - University hospital, Point A Pitre
  - University hospital, Rennes
  - University hospital, Saint-Etienne
  - University hospital, Strasbourg
  - Hospital, Suresnes
  - University hospital, Toulouse
  - Hospital, Valenciennes

IPD SHARING:
Plan to Share IPD: Yes
The French National Data Safety Authority (CNIL) forbids making data freely available without prior agreement. Thus, the data underlying study findings cannot be made freely available because of ethical and legal restrictions. However, individual participant data underlying the results reported in the manuscript (text, tables, figures, and appendices) can be obtained after deidentification. Data can be obtained upon request from the IMPROVE-2 steering committee. Readers may contact: efutier@chu-clermontferrand.fr to request the data.
  The data cannot be freely available for the reasons mentioned above. Data access can be only possible after scientific assessment and data sharing agreement, detailing the type of data requested. This data sharing agreement has to be signed between applicants and the sponsor, Clermont-Ferrand University Hospital.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months following article publication. No end date
Access Criteria: . Data can be obtained upon request from the IMPROVE-2 steering committee. Readers may contact: efutier@chu-clermontferrand.fr to request the data.

REFERENCES:
- [Derived] Futier E, De Jong A, Cirenei C, Godet T, Jabaudon M, Constantin JM, Grillot N, Bouzat P, Henry L, Margetis D, Lebuffe G, Garnier M, Lambert C, Pereira B, Jaber S; IMPROVE-2 Trial investigators. Personalized driving pressure-guided positive end-expiratory pressure in patients at risk of postoperative respiratory failure (IMPROVE-2): a multicenter, pragmatic, randomized clinical trial. Intensive Care Med. 2025 Oct;51(10):1797-1808. doi: 10.1007/s00134-025-08082-x. Epub 2025 Aug 21. PMID 40839096
- [Derived] Khaled L, Godet T, Jaber S, Chanques G, Asehnoune K, Bourdier J, Araujo L, Futier E, Pereira B. Intraoperative protective mechanical ventilation in patients requiring emergency abdominal surgery: the multicentre prospective randomised IMPROVE-2 study protocol. BMJ Open. 2022 May 6;12(5):e054823. doi: 10.1136/bmjopen-2021-054823. PMID 35523498